CLINICAL TRIAL: NCT04459754
Title: Based on the Real World Prospective Cohort Study, Two-way Analysis of the Dominant Population and Corresponding Phenotypic Characteristics of Patients With Colorectal Cancer Treated by Fuzheng Yiliu Therapy Combined With Adjuvant Chemotherapy
Brief Title: Fuzheng Yiliu-1010
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wei Wang, Guangzhou University of Chinese Medicine, The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019KT1089
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer Stage II and III
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuzheng Yiliu group (Experimental)
  Interventions: Drug: Fuzheng Yiliu Formulation
- control group (No Intervention)

INTERVENTIONS:
Drug: Fuzheng Yiliu Formulation — The "prescription for colorectal cancer" Fuzheng Yiliu formulation is a combination of 13 herbal components and it is available in granules form to be dissolved in hot water for consumption.
  Arms: Fuzheng Yiliu group

SUMMARY:
Real world study was used to evaluate the therapeutic effect of Fuzheng anti-tumor therapy on colorectal cancer patients in stage II and III after surgery and standard chemotherapy, and the prediction model of dominant population of Fuzheng anti-tumor therapy was constructed by using real-world data and gene expression profile data.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patients was 18-75 years old;
2. Radical resection of colorectal cancer (negative margin) was performed;
3. Patients with stage II high risk and stage III colorectal cancer confirmed by histology;
4. No liver, peritoneal or distant metastasis was found;
5. Patients with colorectal cancer who received standard chemotherapy or radiotherapy after operation and had no recurrence or metastasis at the end of radiotherapy and chemotherapy;
6. ECoG (Eastern Cooperative Oncology Group) score was 0-1; KPS score was 70 or above;
7. Liver function: SGOT and SGPT were less than 1.5 times of normal value, bilirubin was less than 1.5 mg / dl;
8. Renal function: creatinine < 1.8mg/dl.

Exclusion Criteria:

1. Allergic to the drug of this scheme;
2. Pregnant or lactating women with fertility requirements during the study period;
3. Severe hypertension, coronary heart disease, diabetes and so on, which are under control for half a year due to cardiovascular accident and poor drug control, are accompanied with other uncontrollable benign diseases such as lung, kidney, liver, infection, etc;
4. Participate in other studies before and during treatment;
5. There was a history of other malignant tumors or multi-source tumors within one year;
6. Chronic hepatitis B or C (high copy viral DNA) or activity in HIV infection history or active phase;
7. Patients with tuberculosis or seizures who need to be treated (e.g. steroids or antiepileptic therapy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China